CLINICAL TRIAL: NCT03142919
Title: Response to Inflammatory Challenge in Major Depressive Disorder
Brief Title: Lipopolysaccharide (LPS) Challenge in Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Principal Investigator, Jonathan Savitz, Assistant Professor, Laureate Institute for Brain Research, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2016-002-00
Record Dates: First submitted 2017-04-28; First posted 2017-05-08 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Major Depressive Disorder
Keywords: Mood Disorder; MDD; Endotoxin; MRI; CRP
MeSH Terms: conditions — Depressive Disorder, Major; Mood Disorders | interventions — Lipopolysaccharides; Endotoxins; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- High CRP LPS Intervention (Experimental): High CRP Individuals with Major Depressive Disorder receiving LPS intervention
  Interventions: Biological: Lipopolysaccharide
- Low CRP LPS Intervention (Active Comparator): Low CRP Individuals with Major Depressive Disorder receiving LPS intervention
  Interventions: Biological: Lipopolysaccharide
- High CRP LPS Placebo (Placebo Comparator): High CRP Individuals with Major Depressive Disorder receiving placebo
  Interventions: Biological: Placebo
- Low CRP LPS Placebo (Placebo Comparator): Low CRP Individuals with Major Depressive Disorder receiving placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Lipopolysaccharide — Lipopolysaccharide (LPS) derived from E. Coli group O 113:H10:K negative
  Other Names: Endotoxin, CCRE
  Arms: High CRP LPS Intervention; Low CRP LPS Intervention
Biological: Placebo — Saline solution
  Other Names: Saline solution
  Arms: High CRP LPS Placebo; Low CRP LPS Placebo

SUMMARY:
LPS Challenge in Individuals with Major Depressive Disorder

DETAILED DESCRIPTION:
The aim of this project is to understand the biological differences between two distinct subtypes of depression, patients with and without inflammation as defined by c-reactive protein (CRP). Using a double-blinded, parallel group, placebo-controlled design, participants will be phenotyped before and after a low-dose lipopolysaccharide (LPS) challenge designed to perturb the immune system and trigger a transient, mild inflammatory response. This experimental design will allow for the delineation of the homeostatic mechanisms underlying sensitivity to inflammation-related depression. Low-dose LPS has been used by multiple groups to safely induce transient inflammatory responses in humans.

ELIGIBILITY:
Inclusion Criteria:

Depressed participants will be required to be in good general health (as evaluated during Visit 1, including EKG) and to be 18-55 years of age. Depressed participants will be required to have symptoms of depression (i.e. a PHQ-9 score ≥10) and be unmedicated for at least 3 weeks (8 weeks for fluoxetine) or treated with only one anti-depressant medication. Half the depressed participants (N=50) will be required to have a high-sensitivity C-Reactive Protein (CRP) score of ≥3 mg/L, and half the participants will be required to have a CRP score of ≤1 mg/L.

General Exclusion Criteria:

* Pregnancy
* Previous history of fainting during blood draws.

Medical Conditions:

* A history of a head injury with loss of consciousness.
* Presence of co-morbid medical conditions not limited to but including cardiovascular (e.g., history of acute coronary event, stroke) and neurological diseases (e.g., Parkinson's disease), as well as pain disorders.
* Presence of co-morbid inflammatory disorders such as rheumatoid arthritis or other autoimmune disorders.
* Presence of an uncontrolled medical condition that is deemed by the investigators to interfere with the proposed study procedures, or to put the study participant at undue risk.
* Presence of chronic infection that may elevate pro-inflammatory cytokines.
* Presence of an acute infectious illness or receipt of a vaccination in the two weeks prior to an experimental session.

Psychiatric Disorders:

* Current severe suicidal ideation or attempt within the past 12 months.
* Psychosis
* Bipolar disorder
* Substance abuse or dependence within the previous 6 months
* Age of onset of depression >40 years

Contraindications for MRI:

* Severe claustrophobia
* Bodily implants of unsafe paramagnetic materials such as pace-makers and aneurysm clips.

Medications:

* Current and/or past regular use of hormone-containing medications (excluding contraceptives)
* Current use of non-steroid anti-inflammatory drugs that is deemed by the investigators to potentially confound the results of the study
* Current and/or past regular use of immune modifying drugs that target specific immune responses such as TNF antagonists
* Current use of analgesics such as opioids or history of addiction to opioids or other analgesics
* Current and/or past regular use of cardiovascular medications, including antihypertensive, antiarrhythmic, anti-anginal, and anticoagulant drugs (does not apply where medications are taken for different purpose e.g. anti-hypertensives for migraine).
* Evidence of recreational drug use from urine test.
* Lifetime use of methamphetamine

Health Factors:

* BMI > 35 because of the effects of obesity on pro-inflammatory cytokine activity
* Clinically significant abnormalities on screening laboratory tests
* Abnormal EKG
* In addition, participants who on arrival to the study, show any of the following symptoms will not be allowed to complete the study:

  1. screening supine systolic blood pressure >140 mmHg or <100 mmHg
  2. screening supine diastolic blood pressure >90 mmHg or <60 mmHg
  3. 12-lead EKG demonstrating a PR interval > 0.2 msec, QTc >450 or QRS >120 msec If the QTc exceeds 450 msec, or QRS exceeds 120 msec, the EKG will be repeated 2 more times and the median value will be used
  4. pulse less than 50 beats/minute or greater than 100 beats/minute
  5. temperature greater than 99.5F.

     Non-English speaking participants:
* The majority of the assessments proposed for this study have not been translated from English, thus, non-English speaking volunteers will be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High CRP LPS Intervention | Low CRP LPS Intervention | High CRP LPS Placebo | Low CRP LPS Placebo
Started | 13 | 19 | 13 | 19
Completed | 13 | 19 | 13 | 19
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High CRP LPS Intervention | Low CRP LPS Intervention | High CRP LPS Placebo | Low CRP LPS Placebo | Total
Number analyzed (Participants) | 13 | 19 | 13 | 19 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.0 (11.1) | 30.3 (10.9) | 29.7 (10.0) | 29.6 (10.0) | 31.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 10 | 13 | 47
  Male | 3 | 5 | 3 | 6 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 2
  Asian | 1 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 3 | 2 | 8
  White | 7 | 15 | 9 | 12 | 43
  More than one race | 1 | 2 | 0 | 3 | 6
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Snaith-Hamilton Pleasure Scale [Mean (Standard Deviation); unit: units on a scale] | 27.8 (5.4) | 28.7 (6.3) | 25.7 (4.6) | 26.5 (7.6) | 27.2 (6.2)
Temperature [Median (Inter-Quartile Range); unit: Degrees Fahrenheit] | 97.7 [97.2 to 98.1] | 97.6 [97.2 to 97.8] | 97.3 [97.2 to 97.7] | 97.8 [97.6 to 98.6] | 97.7 [97.3 to 98.1]
Montgomery Asberg Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] | 23.7 (6.5) | 25.1 (5.6) | 22.6 (6.4) | 23.7 (5.7) | 23.9 (5.9)
Interleukin 6 [Median (Inter-Quartile Range); unit: pg/mL] | 0.9 [0.6 to 1.2] | 0.4 [0.3 to 0.6] | 0.5 [0.4 to 0.8] | 0.4 [0.3 to 0.6] | 0.6 [0.4 to 0.8]
Interleukin 10 [Median (Inter-Quartile Range); unit: pg/mL] | 0.2 [0.2 to 0.3] | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.3] | 0.3 [0.1 to 0.4] | 0.2 [0.2 to 0.3]
Tumor Necrosis Factor [Median (Inter-Quartile Range); unit: pg/mL] | 1.8 [1.4 to 2.3] | 1.6 [1.4 to 1.8] | 1.6 [1.5 to 1.8] | 1.5 [1.3 to 2.0] | 1.6 [1.4 to 2.0]

OUTCOME MEASURES:

1. Primary Outcome: Change in Snaith-Hamilton Pleasure Scale (SHAPS)
Description: The SHAPS is a 14-item self-administered questionnaire, with each item scored from 1-4 (strongly agree through strongly disagree; range 14-56), with higher scores indicating greater anticipatory, not consummatory, anhedonia. Disagreement (i.e. score of 3 or 4) on at least three items is defined as indicating clinically significant anhedonia.
Time Frame: 2-hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High CRP LPS Intervention | Low CRP LPS Intervention | High CRP LPS Placebo | Low CRP LPS Placebo
Number analyzed (Participants) | 13 | 19 | 13 | 19
units on a scale | 38.4 (11.3) | 33.2 (8.7) | 27.2 (5.9) | 26.2 (7.0)

2. Secondary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Clinician-administered depression rating scale with scores ranging from 0-60. Higher scores indicate more depression.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High CRP LPS Intervention | Low CRP LPS Intervention | High CRP LPS Placebo | Low CRP LPS Placebo
Number analyzed (Participants) | 13 | 19 | 13 | 19
units on a scale | 9.7 (4.2) | 18.6 (8.6) | 16.0 (9.9) | 18.0 (8.5)

3. Secondary Outcome: Change in Interleukin 6 (IL-6) Protein Levels
Description: pro-inflammatory cytokine measured in pg/mL
Time Frame: 2-hours
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | High CRP LPS Intervention | Low CRP LPS Intervention | High CRP LPS Placebo | Low CRP LPS Placebo
Number analyzed (Participants) | 12 | 13 | 12 | 17
pg/mL | 116.4 [36.2 to 586.9] | 54.0 [20.7 to 152.8] | 0.6 [0.6 to 1.6] | 0.5 [0.3 to 0.6]

4. Secondary Outcome: Change in Interleukin 10 (IL-10) Protein Levels
Description: Measure of systemic inflammation in pg/mL
Time Frame: 2-hours
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | High CRP LPS Intervention | Low CRP LPS Intervention | High CRP LPS Placebo | Low CRP LPS Placebo
Number analyzed (Participants) | 11 | 13 | 11 | 17
pg/mL | 24.1 [17.9 to 34.8] | 12.8 [8.6 to 20.0] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.3]

5. Secondary Outcome: Change in Tumor Necrosis Factor (TNF) Protein Levels
Description: Measure of systemic inflammation in pg/mL
Time Frame: 2-hours
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | High CRP LPS Intervention | Low CRP LPS Intervention | High CRP LPS Placebo | Low CRP LPS Placebo
Number analyzed (Participants) | 11 | 13 | 11 | 17
pg/mL | 146.0 [48.3 to 896.4] | 130.8 [66.7 to 377.4] | 1.5 [1.3 to 2.1] | 1.2 [0.9 to 2.0]

6. Secondary Outcome: Percent Signal Change in Blood Oxygenation Level Dependent Signal (BOLD) of the Ventral Striatum Reward Versus No Reward Condition
Description: Percent change of bold signal in the ventral striatum between conditions p5 and p0 at t2 - % change of bold signal in ventral striatum between conditions p5 and p0 at t1. t1= baseline scan; t2= scan performed 2 hours after LPS/saline. P5= $5 reward; p0=no reward. Data only collected at 2 timepoints.
Time Frame: Baseline line; 2-3 hours
Population: Note that there was missing data for 9 participants
Measure: Mean (Standard Deviation); unit: Percent Signal Change
Groups:
- High CRP LPS VS: High CRP group receiving LPS
- Low CRP LPS: Low CRP group receiving LPS
- Low CRP Saline: Low CRP Group Receiving Saline
- High CRP Saline: High CRP Group Receiving Saline
Arm/Group | High CRP LPS VS | Low CRP LPS | Low CRP Saline | High CRP Saline
Number analyzed (Participants) | 12 | 12 | 18 | 13
Percent Signal Change | -0.09 (0.35) | -0.01 (0.22) | -0.03 (0.21) | 0.01 (0.24)

7. Secondary Outcome: Change in Temperature
Description: Body temperature measured in degrees Fahrenheit.
Time Frame: 4-hours
Measure: Median (Inter-Quartile Range); unit: Degrees Fahrenheit
Arm/Group | High CRP LPS Intervention | Low CRP LPS Intervention | High CRP LPS Placebo | Low CRP LPS Placebo
Number analyzed (Participants) | 13 | 19 | 13 | 19
Degrees Fahrenheit | 98.5 [98.4 to 99.2] | 98.0 [97.6 to 99.2] | 98.1 [97.8 to 98.6] | 98.0 [97.8 to 98.6]

8. Secondary Outcome: Percent Signal Change in Blood Oxygenation Level Dependent Signal (BOLD) of the Insula (Interoceptive vs Exteroceptive Condition)
Description: Percent change of bold signal in the insula between exteroceptive and interoceptive conditions at t2 - % change of bold signal in insula between exteroceptive and interoceptive conditions at t1. t1= baseline scan; t2= scan performed 2 hours after LPS/saline. Data only collected at 2 timepoints.
Time Frame: Baseline line 2-3 hours
Population: Note that there was missing data for 9 participants
Measure: Mean (Standard Deviation); unit: Percent Signal Change
Groups:
- High CRP LPS Insula: High CRP group receiving LPS
Arm/Group | High CRP LPS Insula | Low CRP LPS | Low CRP Saline | High CRP Saline
Number analyzed (Participants) | 12 | 12 | 18 | 13
Percent Signal Change | 0.01 (0.10) | -0.06 (0.15) | 0.01 (0.14) | -0.10 (0.17)

ADVERSE EVENTS:
Time Frame: One week
Arm/Group | High CRP LPS Intervention | Low CRP LPS Intervention | High CRP LPS Placebo | Low CRP LPS Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/19 | 0/13 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/19 | 0/13 | 0/19
Other Adverse Events (participants affected / at risk) | 3/13 | 2/19 | 0/13 | 1/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High CRP LPS Intervention (N=13) | Low CRP LPS Intervention (N=19) | High CRP LPS Placebo (N=13) | Low CRP LPS Placebo (N=19)
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Vasovagal Reaction (General disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Fever (General disorders) | 1 | 0 | 0 | 0
UTI (Infections and infestations) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT03142919/Prot_001.pdf
  • Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT03142919/SAP_003.pdf
  • Informed Consent Form (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT03142919/ICF_000.pdf